CLINICAL TRIAL: NCT01005433
Title: A Dose - Dependent Study of Dexmedetomidine in Suppressing Cardiovascular and Hormonal Responses for Cesarean Delivery
Brief Title: Dexmedetomidine for Cesarean Delivery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King Faisal University (Other)
Responsible Party: Dr. Mohamed R. El-Tahan, King Faisal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10/2009; +966 (56) 9371849
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Pregnant Women Undergoing Cesarean Delivery
Keywords: dexmedetomidine; stress response; cesarean delivery
MeSH Terms: conditions — Fractures, Stress | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dexmedetomidine 0.6 µg/kg/h (Active Comparator): The dexmedetomidine group will receive i.v. infusion of 0.1 mL/kg/h of solution containing 6 µg/mL of dexmedetomidine, at 20 min before induction of anesthesia
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 0.4 µg/kg/h (Active Comparator): The dexmedetomidine group will receive i.v. infusion of 0.1 mL/kg/h of solution containing 4 µg/mL of dexmedetomidine, at 20 min before induction of anesthesia
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 0.2 µg/kg/h (Active Comparator): The dexmedetomidine group will receive i.v. infusion of 0.1 mL/kg/h of solution containing 2 µg/mL of dexmedetomidine, at 20 min before induction of anesthesia.
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): The placebo group (n = 20) will receive an i.v. infusion of 0.1 mL/kg/h saline 0.9%, at 20 min before induction of anesthesia
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — The dexmedetomidine groups (n = 20 for each) will receive i.v. infusion of 0.1 mL/kg/h of solution containing 2, 4, and 6 µg/mL of dexmedetomidine, at 20 min before induction of anesthesia. The placebo and the dexmedetomidine solutions will be looked identical and their infusions will be continued until skin closure, when their infusion rate will be decreased by 50% until 20 min after extubation.
  Arms: Dexmedetomidine 0.2 µg/kg/h; Dexmedetomidine 0.4 µg/kg/h; Dexmedetomidine 0.6 µg/kg/h
Drug: Placebo — The placebo group (n = 20) will receive an i.v. infusion of 0.1 mL/kg/h saline 0.9%, at 30 min before induction of anesthesia. The placebo solution will be looked identical and their infusions will be continued until skin closure, when the infusion rate will be decreased by 50% until 20 min after extubation. The test solution will be prepared by one anesthesiologist before induction of anesthesia.
  Arms: Placebo

SUMMARY:
Regional anesthesia has become the anesthetic of choice for cesarean section in most countries; however, some women still prefer general anesthesia techniques. There are many trials for the pharmacological modifications of the sympathetic response to surgery, including opioids, tenoxicam, ketorolac, lidocaine and paracetamol. However, opioid administration to the mother before delivery has adverse neonatal effects. This research is a novel trial on the use of dexmedetomidine for suppression of the hemodynamic and hormonal responses of cesarean delivery.

DETAILED DESCRIPTION:
Literature Review Regional anesthesia has become the anesthetic of choice for cesarean section in most countries; however, some women still prefer general anesthesia rather than regional techniques. There are many published controlled trials for the pharmacological modifications of the sympathetic response to laryngoscopy, tracheal intubation, and surgical stimulation, including opioids, tenoxicam, ketorolac, lidocaine and paracetamol.1-6 However, opioid administration to the mother before delivery has adverse neonatal respiratory depression.1

Dexmedetomidine, a specific [alpha]2-adrenoceptor agonist, has been approved for clinical use for sedation of patients who need mechanical ventilation in the intensive care unit. 7 It has shown sedative, analgesic, and anxiolytic effects after intravenous (IV) administration.8It is felt that the sedative effect of dexmedetomidine is safe and suited for extubation under sedation because it has little effect on respiration.9

An older study tested the effects of preoperative administration of dexmedetomidine 10 min prior to the induction of anesthesia on hemodynamic changes after intubation in 96 women undergoing abdominal hysterectomy. They found that the increase in blood pressure and heart rate was significantly less in the higher dexmedetomidine (0.6 µg/kg) group than in the saline group (P < 0.01). Also, the postintubation increase in heart rate was significantly less (P < 0.05) with the use of dexmedetomidine 0.6 µg/kg (increase of 18 ± 3 bpm) compared to fentanyl (increase of 26 ± 3 bpm). In patients receiving dexmedetomidine 0.3 µg/kg, the increase in blood pressure or heart rate did not differ from those receiving saline.10

Others found that a single pre-induction intravenous dose of dexmedetomidine 2 µg/kg in 50 patients undergoing minor orthopaedic and general surgery was associated with reduced the hemodynamic response to tracheal intubation and extubation, intra-operative heart rate variability, postoperative analgesic and anti-emetic requirements and lower peri-operative serum catecholamine concentrations. However, there were more frequent episodes of hypotension and bradycardia.11

Similarly, others reported that preoperative administration of a single dose of dexmedetomidine 50 patients scheduled for elective minor surgery resulted in progressive increases in sedation, blunted the haemodynamic responses during laryngoscopy, and reduced opioid and anaesthetic requirements. 12

Recently, others found that a single dose of 0.5 µg/kg dexmedetomidine given before induction of anesthesia in 40 ASA physical status I and II patients, aged 20 to 60 years, who were scheduled for elective cholecystectomy, decreased thiopental requirements, lower heart rate values, minimal effects on ejection fraction (EF), end-diastolic index (EDI), cardiac index (CI), and stroke volume index (SVI), or any effect on recovery time.13

Esmaoglu and co'workers compared the use of midazolam loading dose of 0.05 mg/kg followed by an infusion of 0.1 mg/kg/h and dexmedetomidine loading dose 1 µg/kg per 20 minutes, followed by continuous infusion at 0.7 µg/kg/h in 40 women with eclampsia requiring termination of pregnancy by caesarean delivery in intensive care unit (ICU). They concluded that dexmedetomidine sedation in eclampsia patients is effective in reducing the demand for antihypertensive medicine and duration of ICU stay.14

The safety of the use of dexmedetomidine on neonatal outcome is a very important issue. Experimental study on acute exposure of rats to dexmedetomidine at the anticipated delivery time recorded absence of any adverse effects on perinatal morphology of pups, their birth weight, crown-rump length, physical growth and postnatal behavioural performances.15 Others studied the transfer of clonidine and dexmedetomidine across the isolated perfused human placenta. Dexmedetomidine disappeared faster than clonidine from the maternal circulation, while even less dexmedetomidine was transported into the fetal circulation. This was due to its greater placental tissue retention, the basis for which probably is the higher lipophilicity of dexmedetomidine.16

There are many published reports about the safety use of dexmedetomidine in neonates and infants. Some authors described the successful use of dexmedetomidine as the sole anesthetic for four infants requiring general anesthesia for direct laryngoscopy and bronchoscopy with spontaneous ventilation with adequate surgical conditions and the hemodynamic and respiratory profiles.17-18 Others suggested that invasive procedures can be successfully performed in spontaneously breathing infants and toddlers with congenital heart disease using dexmedetomidine 1-3 µg/kg alone or in combination with low dose ketamine.19Others reported a case of an infant undergoing endoscopic repair of a laryngeal cleft where the combination of dexmedetomidine and propofol infusions was successfully used as the anesthetic technique.

There is currently no FDA-approved usage in children. Despite this fact, there are more than 1,000 pediatric-aged patients reported in the literature who have received dexmedetomidine for a variety of clinical applications in and out of the operating room. 20

Recently, there is a published interested case report about the successful use of dexmedetomidine 1 µg/kg followed with 1 µg/kg/h for 10 minutes before cesarean delivery to facilitate awake fiberoptic endotracheal intubation patient with spinal muscular atrophy type III with provided adequate sedation, without respiratory compromise. Although pharmacokinetic data cannot be determined, this case confirms existing in vitro data that dexmedetomidine has significant placental transfer. Nevertheless, serious neonatal effects were not detected.21 Similarly, others used, i.v. dexmedetomidine successfully as an adjunct to opioid-based PCA and general anesthesia for the respective provision of labor analgesia and cesarean delivery anesthesia in a parturient with a tethered spinal cord, with favourable maternal and neonatal outcome.22

There is an interested editorial report summarized that the practitioners of obstetric analgesia would probably appreciate an additional agent for the provision of pain relief for parturients who are unable or unwilling to receive neuraxial block. The role of low-dose infusion of dexmedetomidine to maintain light sedation and haemodynamic stability with minimal risk of respiratory depression could be advantageous, especially with proper patient selection and monitoring. Its effects on the pregnant uterus, utero-placental unit and the neonate must be rigorously examined.23

Project Objectives:

We hypothesize that the the preoperative use of different doses of i.v. dexmedetomidine , namely 0.2, 0.4 and 0.6 µg/kg/h from the preanesthesia period to the postoperative period for uncomplicated cesarean delivery would reduce the maternal hemodynamic and hormonal responses to endotracheal intubation, surgical stimulation and extubation with improved quality of postoperative analgesia without harmful neonatal effects.

The aims of the present study are:

Our research efforts will focus on identifying the effects of 0.2, 0.4 and 0.6 µg/kg/h dexmedetomidine for uncomplicated cesarean delivery on the followings.

1. Hemodynamic [heart rate, systolic and mean blood pressure] changes.
2. The perioperative changes in plasma cortisol concentrations.
3. The perioperative changes in plasma catecholamines concentrations, namely, epinephrine and norepinephrine.
4. The neonatal outcome as regarding Apgar score, the neurologic and adaptive capacity score (NACS), and umbilical cord venous and arterial blood gases analyses.
5. The quality of extubation conditions.
6. The quality of postoperative analgesia.
7. The incidence of the major complications (respiratory, cardiovascular events, and neonatal adverse outcome).

Project Design:

Study Design:

This prospective randomized placebo-controlled double-blinded study will be carried out from at the Maternity Unit - King Fahd University Hospital, after approval of the Local Institutional Ethical Committee.

Study Phases: The project comprised of five phases as follow:

• Phase I: Literature review collection and writing which will spend 1 months.

• Phase II: Pilot Study for 1 months to determine the sample size required to detect significant changes [Alpha error 0.05] in the hemodynamic responses [heart rate and blood pressure] to intubation, surgical stimulation and extubation with the preoperative use of dexmedetomidine for uncomplicated cesarean delivery to achieve an 85% power for that study.

• Phase III: (7 months) A. To test the primary effects of the preoperative use of different doses of dexmedetomidine [0.2, 0.4 and 0.6 µg/kg/h] for uncomplicated cesarean delivery: on perioperative hemodynamic responses, cortisol, epinephrine and norepinephrine changes B. To test the secondary outcome variables included; the neonatal outcome as regarding Apgar score, the neurologic and adaptive capacity score (NACS), and umbilical cord venous and arterial blood gases analyses, the quality of extubation conditions and postoperative analgesia and the incidence of the major complications (respiratory, cardiovascular events, and neonatal adverse outcome).

Sampling Site:

The study will be conducted in the DR suite and maternity unit at the King Fahd Hospital of the University - Al khobar Study period: For 9 months. I. Patient Selection: patients aged 18-60 years (ASA physical status II-III) scheduled for elective in about 80 women (American Society of Anesthesiologists [ASA] I and II), with uncomplicated, singleton pregnancies of at least 36 weeks' gestation, who will receive regional anesthesia and were scheduled for elective cesarean delivery under general anesthesia. We will exclude women with a history of cardiac, liver, or kidney diseases; allergy to amide local anesthetics; epilepsy; those taking cardiovascular medications; and those with pregnancy-induced hypertension, evidence of intrauterine growth restriction, or fetal compromise.

I. Patient Groups and Study Protocol: All patients will be randomly assigned using sealed envelopes included the computer generated randomized code into four groups; to receive either placebo (saline) [group 1], dexmedetomidine [0.2, 0.4 and 0.6 µg/kg/h in groups 2, 3, and 4 respectively, will started 10 minutes before induction of general anesthesia

II. Anesthesia and Surgery:

All parturients will receive oral ranitidine 150 mg on the night before and on the morning of surgery and 30 mL of 0.3 mol/L sodium citrate 15 min before induction. Lactated Ringer's solution (500 mL) will infused over 20 min. Left uterine displacement will be maintained before induction.

The subjects will be allocated randomly to two groups,using a computer-generated randomization code. The placebo group (n = 20) will receive an i.v. infusion of 0.1 mL/kg/h saline 0.9%, at 20 min before induction of anesthesia. The dexmedetomidine groups (n = 20 for each) will receive i.v. infusion of 0.1 mL/kg/h of solution containing 2, 4, and 6 µg/mL of dexmedetomidine, at 20 min before induction of anesthesia. The placebo and the dexmedetomidine solutions will be looked identical and their infusions will be continued until skin closure, when their infusion rate will be decreased by 50% until 20 min after extubation. The test solution will be prepared by one anesthesiologist before induction of anesthesia. Another anesthesiologist, who will be blinded to the study solution, will give the anesthetic and will perform the assessments. All staff in the operating room will be unaware of the randomization code.

Maternal monitoring will include electrocardiography, noninvasive blood pressure, pulse oximetry, end-tidal sevoflurane and carbon dioxide (EtCO2) concentrations, neuromuscular blockade, and response entropy (RE) and state entropy (SE) using the Datex-Ohmeda S/5 Entropy Module (M-EntropyTM) (Datex-Ohmeda Division, Instrumentarium Corporation, Helsinki, Finland).. After preoxygenation for 5 min, a rapid-sequence induction will be performed with propofol 1.5-2.5 mg/kg and suxamethonium 1.5 mg/kg. Cricoid pressure will be applied, laryngoscopy will be performed after the 1-min blood pressure recording, and tracheal intubation will be completed before the 2-min reading. Anesthesia will be maintained with a 45% of oxygen with 0.5-1 MAC of sevoflurane based on entropy reading where the end-point was SE 50 and SE-RE difference less than 10. Rocuronium 0.6 mg/kg will be given for muscle relaxation to maintain suppression of the second twitch using a train-of-four stimulation.

. The patients'lungs will be ventilated to maintain an EtCO2 of 4-4.6 kPa. After the umbilical cord will be clamped, infusions of 10 U oxytocin and fentanyl 2 μg/kg will be given. Sevoflurane will be discontinued and study drug infusion rate will be decreased by 50% at the start of skin closure. At the end of surgery, residual neuromuscular block will be antagonized with neostigmine 50 μg/kg and atropine 20 μg/kg, and the trachea will be extubated. The study drug infusion will be discontinued 20 min after extubation.

III. The Investigators who will be involved with subsequent postoperative patient assessment will be blinded of the patient group.

IV. Clinical Examination: will include times for induction to delivery (I-D), extubation (time from discontinuation of sevoflurane to extubation), and spontaneous ventilation (time between beginning of spontaneous breathing and extubation) will be recorded. The quality of tracheal extubation will be was evaluated using a 5-point rating scale: 1, no coughing or straining; 2, very smooth, minimal coughing; 3, moderate coughing; 4, marked coughing or straining; and 5, poor extubation, very uncomfortable.25 Heart rate and mean arterial pressure (MAP) will be recorded before and 15 min after bolus infusion; at 1, 2, 3, 4, 5, 6, 7, 8, 9, and 10 min after induction; 15 and 30 min after delivery; and 0, 1, 5, 15, 30, and 60 min after extubation.

The obstetrician will be assessed uterine tone by palpation every 5 min after delivery of the placenta, using a 10-cm visual analogue score (VAS; 0, well contracted; 10, completely relaxed). If uterine tone remained unsatisfactory after 3 min, an additional 5-U bolus of oxytocin will be administered.

All neonates will be assessed by a pediatrician unaware of the mothers' randomization. Apgar scores at 1 and 5 min, and newborns' blood pressure, heart rate, temperature, arterial oxygen saturation, and the neurologic and adaptive capacity score (NACS) will be recorded at 15 min and at 2 and 24 h after delivery. NACS gives a total score: the maximum is 40, and a score of 35-40 denotes vigor.26 The percentages of infants scoring 35 or less will be determined.

The presence of perioperative side effects, including bradyarrhythmia, hypotension, sedation, nausea and vomiting, neonatal hypothermia, bradycardia or respiratory depression will be reported.

V. Blood Biochemistry: will include the neonatal umbilical artery (UA) and umbilical vein (UV) samples collection from a double-clamped segment of umbilical cord for the measurement of blood pH, gas tensions, and base excess.

VI. Samples Collection and Analysis For the hormonal assays: Maternal venous blood samples (MV) will be collected for assay of cortisol, epinephrine and norepinephrine concentrations, at five points: preoperatively, immediately after bolus infusion, 5 min after intubation, 1 h after delivery, and 1 h after continuous infusion.

1. . Type of samples: centrifuged stored aliquots of serum at -70°C.
2. . Laboratory Analysis:

   1. Plasma cortisol levels will be determined using a radioimmunoassay technique (Gamma Coat Cortisol 125IRIA; Nihon Sheering, Chiba, Japan).
   2. Plasma catecholamines [epinephrine and norepinephrine] levels will be determined using a radioimmunoassay technique.

IV. Statistical Analysis: 1month Statistical analysis will be performed using the Statistical Package for the Social Sciences (SPSS Inc., Chicago, IL). Data will be tested for normality using the Kolmogorov-Smirnov test. Repeated-measures analysis of variance will be used for analysis of serial changes in the hemodynamic data at different times after administration of dexmedetomidine . Chi-square test will be used for categorical data. Parametric variables will be analyzed by one way ANOVA comparisons among the four groups and will be followed by the post hoc Tukey's HSD (honestly significant difference) test. The Kruskal-Wallis one-way ANOVA will be performed for intergroup comparisons for the non-parametric hormonal values and post hoc pairwise comparisons will be done using the Wilcoxon rank sum t test. Data will be expressed as mean (SD), number (%), or median [range]. A value of p < 0.05 will be considered to represent statistical significance.

V.Report Writing:2 months

ELIGIBILITY:
Inclusion Criteria:

* 80 women aged 18-45 years (ASA physical status II-III)with uncomplicated, singleton pregnancies of at least 36 weeks' gestation scheduled for elective cesarean delivery under general anesthesia.

Exclusion Criteria:

* women with a history of cardiac, liver, or kidney diseases;
* women with allergy to amide local anesthetics;
* women with epilepsy;
* those taking cardiovascular medications;
* those with pregnancy-induced hypertension;
* women with evidence of intrauterine growth restriction or fetal compromise.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
identifying the effects of 0.2, 0.4 and 0.6 µg/kg/h dexmedetomidine for on 1. Hemodynamic [heart rate, systolic and mean blood pressure] changes. 2. The perioperative changes in plasma cortisol and catecholamines concentrations | before and 15 min after infusion; each 1 min for 10 min after induction; 15 and 30 min after delivery; and 0, 1, 5, 15, 30, and 60 min after extubation

SECONDARY OUTCOMES:
Apgar score, the neurologic and adaptive capacity score (NACS), and umbilical cord venous and arterial blood gases analyses.The quality of extubation and analgesia.major complications (respiratory, cardiovascular events, and neonatal adverse outcome | after delivery, and postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R El Tahan, M.D, Principal Investigator — King Faisal University
Locations (1):
- King Faisal University, Dammam, Eastern Province, Saudi Arabia